CLINICAL TRIAL: NCT05894018
Title: A Phase II Clinical Trial Evaluating the Safety and Efficacy of Radioactive Particle and Fluzoparib Combination Therapy in the Treatment of Advanced Unresectable Soft Tissue Sarcoma
Brief Title: Brachytherapy (Iodine-125 Seeds) and Fluzoparib Combination Therapy for Advanced Unresectable Soft Tissue Sarcoma
Acronym: RAFAS-001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujun Zhang (Other)
Responsible Party: Sponsor-Investigator, Fujun Zhang, Prof., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2023-135-02
Record Dates: First submitted 2023-05-26; First posted 2023-06-08 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Sarcoma,Soft Tissue; Brachytherapy; Poly(ADP-ribose) Polymerase Inhibitors
Keywords: Fluzoparib; Radioactive particles; Iodine-125 seed
MeSH Terms: conditions — Sarcoma | interventions — fluzoparib

STUDY DESIGN:
Intervention Model Description: Fluzoparib 150 mg Bid was given orally after meals for 2 months (60 days) in a continuous cycle 48 h after radioactive particle implantation. The maximum cumulative dosing period is 1 year. Tumor assessment was performed in each cycle. The first cycle is evaluated every month. Patients in partial remission (PR) or patients with stable disease (SD) will be supplemented with additional particle implantations (≤3) according to the dose prescribed by the physician, noting the need to discontinue the drug for at least 5 days prior to surgery and to continue oral Fluzoparib for 2 days after surgery until 6 months after the last particle implantation. Patients with intolerable toxicity or patient requested discontinuation or disease progression (PD) were withdrawn from the trial and entered into survival follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib+radioactive particle implantation (Experimental): Fluzoparib 150 mg bid was given orally after meals for 2 months (60 days) in a continuous cycle 48h after radioactive particle implantation.
  Interventions: Drug: Fluzoparib; Procedure: Radioactive particle implantation

INTERVENTIONS:
Drug: Fluzoparib — 150mg, orally, bid
Procedure: Radioactive particle implantation — Radioactive iodine-125 seeds implantation

SUMMARY:
To evaluate the effectiveness and safety of radioactive particles in combination with the PARP inhibitor fluzoparib in the treatment of advanced inoperable soft tissue sarcoma.

DETAILED DESCRIPTION:
Fluzoparib 150 mg Bid was given orally after meals for 2 months (60 days) in a continuous cycle 48 h after radioactive particle implantation. The maximum cumulative dosing period is 1 year. Tumor assessment was performed in each cycle. The first cycle is evaluated every month. Patients in partial remission (PR) or patients with stable disease (SD) will be supplemented with additional particle implantations (≤3) according to the dose prescribed by the physician, noting the need to discontinue the drug for at least 5 days prior to surgery and to continue oral Fluzoparib for 2 days after surgery until 6 months after the last particle implantation. Patients with intolerable toxicity or patient requested discontinuation or disease progression (PD) were withdrawn from the trial and entered into survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate in this study and sign an informed consent form;
2. Age ≥18 (calculated on the day of signing the informed consent), regardless of gender;
3. Pathologically confirmed soft tissue sarcoma, with at least one measurable lesion according to RECIST 1.1 criteria on CT or MRI scan, within 28 days before the first study treatment (the longest diameter of the lesion ≥10 mm or the short diameter of swollen lymph node ≥15 mm);
4. A single lesion ≤5cm and no more than 5 lesions;
5. Received systemic therapy (such as standard treatment: doxorubicin plus ifosfamide) ± surgical resection as the first-line treatment;
6. Able to swallow pills normally;
7. ECOG performance status of 0-1;
8. Expected survival period ≥12 weeks;
9. Normal function of important organs, including:

Absolute neutrophil count ≥1.5×109/L;Platelets ≥80×109/L;Hemoglobin ≥90 g/L;Serum albumin ≥28 g/L;Thyroid-stimulating hormone (TSH) ≤1×ULN (if abnormal, FT3 and FT4 levels should be examined simultaneously, and if FT3 and FT4 levels are normal, patients can be included);Bilirubin ≤1.5×ULN (within 7 days before the first treatment);ALT and AST ≤3×ULN (within 7 days before the first treatment);Alkaline phosphatase (AKP) ≤2.5×ULN;Serum creatinine ≤1.5×ULN; Non-surgically sterilized or fertile female patients need to use a medically recognized contraceptive measure (such as an intrauterine device, birth control pills, or condoms) during the study treatment period and within 3 months after the end of the study treatment. Fertile female patients who are not surgically sterilized must have a negative serum or urine HCG test within 72 hours before study enrollment and must not be breastfeeding. Male patients with fertile female partners should also use effective contraception during the trial period and for 3 months after the last dose of the study treatment.

Exclusion Criteria:

1. Clinical cardiac symptoms or disease that were not well controlled, such as: NYHA class 2 or higher heart failure, unstable angina, myocardial infarction within 1 year, clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention, QTc>450ms (men); QTc>470ms (women);
2. Coagulation abnormal function (INR>2.0, PT>16s), bleeding tendency or on thrombolytic or anticoagulant therapy, prophylactic use of low-dose aspirin, low-molecular heparin allowed;
3. Clinically significant bleeding symptoms or clear bleeding tendency within 3 months prior to enrollment, such as daily cough/hemoptysis of 2.5 ml or more, gastrointestinal bleeding, esophagogastric fundic varices with bleeding risk ;
4. Arterial/venous thrombotic events such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, and cerebrovascular disease) that occurred within 6 months prior to enrollment. ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
5. Known hereditary or acquired bleeding and thrombotic predisposition (e.g., hemophiliacs, coagulation disorders, thrombocytopenia, etc.);
6. Patients who have received prior chemotherapy, surgery, less than 4 weeks after completion of treatment (last dose) and prior to study dosing; or patients who have not recovered from adverse events (other than alopecia) caused by prior treatment to ≤ CTCAE grade 1;
7. Patients with active infection, unexplained fever ≥38.5°C within 7 days prior to dosing, or white blood cell count >15×109/L at baseline;
8. Patients with other malignancies (except cured basal cell carcinoma of the skin and cervical carcinoma in situ) within the previous 3 years or concurrently;
9. Patients with established bone metastases who have received, within 4 weeks prior to enrollment in the study;
10. Prior external radiotherapy to the lesion;
11. Pregnant or breastfeeding women, or women of childbearing age who do not wish to use contraception;
12. Patients who, in the judgment of the investigator, have other factors that may affect the outcome of the study or force the termination of the study, such as alcoholism, substance abuse, other serious illnesses (including mental illness) requiring comorbid treatment, severe abnormal laboratory tests, accompanied by family or social factors that would affect the safety of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 12 months
  ORR was defined as the percentage of participants with a best overall response of The proportion of patients achieving complete response (CR, tumor disappearance) or partial response (PR, tumor shrinkage) as evaluated by researchers based on the RECIST 1.1 criteria after receiving treatment.

SECONDARY OUTCOMES:
Progression-free survival rate(PFS) | 6 months
  Based on RECIST 1.1 criteria, all patients were evaluated from the first day of iodine-125 seeds brachytherapy treatment until objective tumor progression or death from any cause. The percentage of subjects with progression-free survival at 6 months after treatment was calculated using the Kaplan-Meier method.
Progression-free survival rate(PFS) | 12 months
  Based on RECIST 1.1 criteria, all patients were evaluated from the first day of iodine-125 seeds brachytherapy treatment until objective tumor progression or death from any cause. The percentage of subjects with progression-free survival at 12 months after treatment was calculated using the Kaplan-Meier method.
Progression-free survival rate(PFS) | 18 months
  Based on RECIST 1.1 criteria, all patients were evaluated from the first day of iodine-125 seeds brachytherapy treatment until objective tumor progression or death from any cause. The percentage of subjects with progression-free survival at 18 months after treatment was calculated using the Kaplan-Meier method.
Disease control rate(DCR) | 12 months
  Defined as the proportion of subjects achieving complete response (CR), partial response (PR), or stable disease (SD) for at least 4 weeks after treatment.
Overall survival(OS) | 12 months
  Defined as the time interval from the date of enrollment to death from any cause, with censoring at the last known alive date if no death has occurred.
Overall survival rate | 6 months
  Defined as the proportion of patients who are still alive at 6 months from the initiation of treatment during follow-up.
Overall survival rate | 12 months
  Defined as the proportion of patients who are still alive at 12 months from the initiation of treatment during follow-up.
Overall survival rate | 18 months
  Defined as the proportion of patients who are still alive at 18 months from the initiation
AE, SAE | 12 months
  The incidence of adverse events (AE), serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Fujun Zhang, Ph.D,M.D, Study Director — Sun Yat-sen University; Xing Zhang, Ph.D,M.D, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No